CLINICAL TRIAL: NCT01285453
Title: A Safety, Tolerability Study of Intravenous ASA404 Administered in Combination With Docetaxel in Japanese Patients With Advanced or Recurrent Solid Tumors
Brief Title: Safety and Tolerability of ASA404 Administered in Combination With Docetaxel in Japanese Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASA404A1102
Record Dates: First submitted 2011-01-26; First posted 2011-01-28 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2012-11

CONDITIONS: Advanced or Recurrent Solid Tumors
Keywords: ASA404,; vadimezan,; docetaxel
MeSH Terms: interventions — vadimezan

ARMS (1):
- ASA404 (Experimental)
  Interventions: Drug: vadimezan

INTERVENTIONS:
Drug: vadimezan
  Other Names: ASA404

SUMMARY:
This study will assess the tolerability of combination therapy with ASA404 and docetaxel in Japanese patients with advanced or recurrent solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed solid tumors whose disease has progressed or recurred after treatment at lease one therapy, except docetaxel
2. WHO Performance Status of 0-1

Exclusion Criteria:

1. Patients having symptomatic CNS tumor/metastasis and requiring treatment
2. Patients who have received prior therapy with ASA404 or other vascular disrupting agents
3. Patients with systolic BP > 160mmHg and/or diastolic BP > 90mmHg
4. Patients with fluid retention
5. Patients with any one of cardiotoxicities
6. Concomitant use of drugs with a risk of prolonging the QT interval
7. Known allergy or hypersensitivity to taxane or polysorbate 80

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Japan (2):
  - Novartis Investigative Site, Aichi
  - Novartis Investigative Site, Osaka

REFERENCES:
- [Derived] Daga H, Hida T, Ishikawa S, Shimizu J, Tokunaga S, Horio Y, Kobayashi K, Takeda K. The safety and tolerability of intravenous ASA404 when administered in combination with docetaxel (60 or 75 mg/m(2)) in Japanese patients with advanced or recurrent solid tumors. Jpn J Clin Oncol. 2011 Sep;41(9):1067-73. doi: 10.1093/jjco/hyr110. Epub 2011 Aug 10. PMID 21835825
- See also: Results for CASA404A1102 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4003